CLINICAL TRIAL: NCT00172159
Title: Influence of Neoadjuvant Therapy on the Resectability of Hepatic Metastases From Colorectal Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 170CL6
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2000-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Chemotherapy; Surgery; Liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Procedure: Hepatic resection

SUMMARY:
More and more colorectal surgeons believe that surgical resections of hepatic metastases from colorectal cancer is the only chance for cure of patients. The five-year survival for patients with hepatic metastasis from colorectal cancer after surgical resection is approximately 30 %. However, most hepatic metastases from colorectal cancer were inoperable. With the progress of chemotherapy, for example, the combination of the 5-Fu, leucovorin, and oxaliplatin, some surgeons advocated that approximately 20% of inoperable liver metastases will be converted to operable case, thus providing the long-term survival for patients. In this study, we made a phase Ⅱ clinical trial regarding the use of the Folfox-4 regimens in the neo-adjuvant treatment of inoperable hepatic metastases. Our aims is to evaluate the tumor response rate for this regimen, the rate of resectability of liver metastases, progression free survival and overall survival of patients. In addition, the difference between the reports from Western and Oriental countries will be analyzed. We believe this study will provide new perspectives regarding the most beneficial treatment modalities for the patients with hepatic metastases from colorectal cancer.

DETAILED DESCRIPTION:
More and more colorectal surgeons believe that surgical resections of hepatic metastases from colorectal cancer is the only chance for cure of patients. The five-year survival for patients with hepatic metastasis from colorectal cancer after surgical resection is approximately 30 %. However, most hepatic metastases from colorectal cancer were inoperable. With the progress of chemotherapy, for example, the combination of the 5-Fu, leucovorin, and oxaliplatin, some surgeons advocated that approximately 20% of inoperable liver metastases will be converted to operable case, thus providing the long-term survival for patients. In this study, we made a phase Ⅱ clinical trial regarding the use of the Folfox-4 regimens in the neo-adjuvant treatment of inoperable hepatic metastases. Our aims is to evaluate the tumor response rate for this regimen, the rate of resectability of liver metastases, progression free survival and overall survival of patients. In addition, the difference between the reports from Western and Oriental countries will be analyzed. We believe this study will provide new perspectives regarding the most beneficial treatment modalities for the patients with hepatic metastases from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. colorectal cancer with primarily non-resectable hepatic metastasis, defined as (one of the following): (1) liver metastases > five; (2) liver metastases are anatomically or functionally non-resectable (e.g. insufficient functional liver tissue, liver venous infiltration, liver arterial infiltration, …..) 2. No extra-hepatic disease 3. No prior chemotherapy, except adjuvant chemotherapy 4. Primary tumor resection >1 month 5. Signed written informed consent 6. Male or female 18 - 75 years of age 7. Histologically confirmed adenocarcinoma of the colon or rectum 8. No extra-hepatic disease 9. Presence of at least one bi-dimensional indicator lesion measurable by CT scan or MRI not in an irradiated area 10. Life expectancy of >= 3 months 11. Karnofsky performance status >= 70% 12. Neutrophils >= 1.5 x 109/L, platelets >= 100 x 109/L, and hemoglobin >= 9 g/dL 13. Bilirubin level < 1.5 x ULN 14. ASAT and ALAT £ 2.5 x ULN (<= 5 x ULN if liver metastasis are present) 15 Serum creatinine < 1.5 x ULN 16. Effective contraception for both male and female patients if the risk of conception exists

Exclusion Criteria:

* 1. Brain metastasis (known or suspected) 2. Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol 3. Any investigational agent(s) within 4 weeks prior to entry 4. Previous exposure to monoclonal antibodies, signal transduction inhibitors or other EGFR-targeting therapy 5. Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months 6. Acute or subacute intestinal occlusion or history of inflammatory bowel disease Known grade 3 or 4 allergic reaction to any of the components of the treatment 7. Known drug abuse/ alcohol abuse 8. Legal incapacity or limited legal capacity 9. Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent 10. Women who are pregnant or breastfeeding 11. Clinically relevant peripheral neuropathy 12. Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for >= 5 years will be allowed to enter the trial)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Study Completion 2005-06 (Estimated)

PRIMARY OUTCOMES:
Response rate and resectability after neoadjuvant therapy.

SECONDARY OUTCOMES:
Survival of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung Liang, M.D., Ph.D., Principal Investigator — Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C.
Locations (1):
- Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C., Taipei, Taiwan